CLINICAL TRIAL: NCT06007339
Title: Safety and Performance Study for Venous Large Hole Vascular Closure Device - ELITE Study
Brief Title: PerQseal® Elite Venous Clinical Study (ELITE-Venous)
Acronym: ELITE-Venous
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vivasure Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P934-00
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Large Hole Percutaneous Venous Closure
Keywords: Venous Closure; Percutaneous closure; Large bore closure

STUDY DESIGN:
Intervention Model Description: This study is a prospective, multicentre, single-arm study to investigate the safety and efficacy of the PerQseal Elite.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational Device Arm (PerQseal Elite- Venous) (Experimental): Large hole percutaneous venous closure device - PerQseal Elite
  Interventions: Device: PerQseal ELITE

INTERVENTIONS:
Device: PerQseal ELITE — The term PerQseal Elite used singularly refers to the closure system comprising the closure device and Introducer. These individually are referred to as: "PerQseal Elite VCD" or "PerQseal Elite closure device" and/or "PerQseal Elite Introducer".
  Other Names: Percutaneous ELITE Venous Closure Device

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the PerQseal Elite vascular closure system when used to achieve haemostasis of common femoral venotomies created by 14 to 22F sheaths (venotomy up to 26F) in patients undergoing percutaneous catheter-based interventional procedures, with sufficient rigor to provide robust scientific evidence for the demonstration of clinical safety and efficacy of the PerQseal Elite closure system to support a CE-mark and a PMA submission.

DETAILED DESCRIPTION:
This study is a prospective, multicentre, single-arm study to investigate the safety and efficacy of the PerQseal Elite in up to 97 patients at up to 12 European investigational sites. The study shall not be blinded prior to, during or post the procedure. Patients undergoing a percutaneous catheter-based venous interventional procedure (e.g., mitral valve repair, leadless pacemaker implantation, circulatory assist or ECMO via large bore femoral vein catheter) requiring a venotomy created by 14 to 22F sheaths (venotomies up to 26F), via the common femoral vein will be screened against the study inclusion/exclusion criteria.

All subjects shall have a 30-minute, 60-minute, pre-discharge (~48 hours), 30-Days ± 7-Days and 180-Days ± 30-Days follow-up assessments.

All safety data from the study will be assessed by the Data Safety Monitoring Committee on a continuous basis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years.
2. Clinically indicated for a percutaneous venous interventional catheter-based procedure, e.g., mitral valve edge to edge repair, left atrial appendage device closure, leadless pacemaker implantation, patent foramen ovale closure or use of a circulatory assist device or extracorporeal oxygenation using a common femoral venotomy created by a 14 to 22F sheath (venotomy up to 26F).
3. Subject is willing and able to provide appropriate study-specific informed consent, follow protocol procedures, and comply with follow-up visit requirements.
4. Females who are not pregnant or lactating and not planning to become pregnant for the duration of the study.

Baseline Exclusion Criteria:

1. Evidence of current systemic bacterial or cutaneous infection, including groin infection,
2. Known bleeding diathesis, unstable INR, definite or potential coagulopathy, platelet count < 100,000/μl or subjects on long term anticoagulants with an INR > 2.2 within 12 hours prior to index procedure,
3. Significant anaemia (example: haemoglobin < 8 g/dL or haematocrit < 22%), within 24 hours prior to index procedure,
4. Known type II heparin-induced thrombocytopenia,
5. Documented right ventricular dysfunction < 13%,
6. Ipsilateral or contralateral lower extremity amputation,
7. Previous groin surgery within the region of the ipsilateral vessel access,
8. Common femoral vein diameter stenosis > 50% or previous bypass surgery/stent placement in the common femoral vein of target leg,
9. Known existing nerve damage in the target leg,
10. Nephrotic syndrome or renal insufficiency (Glomerular Filtration Rate ≤ 30 ml/min or baseline serum creatinine > 2.5 mg/dl) or on renal replacement therapy or albumin level < 3.5 g/dl or symptoms of pitting oedema,
11. Systolic pulmonary artery pressure > 60 mmHg
12. Known allergy to any of the materials used in the PerQseal Elite device (refer to Investigator's Brochure),
13. Subject is unsuitable for surgical repair of the target leg access site,
14. Subject has undergone a percutaneous procedure greater than 8F sheath in the target vessel, within the 90-days prior to index procedure,
15. Subject has undergone a percutaneous procedure of 8F sheath or less using an absorbable intravascular closure device for haemostasis, in the target vessel, within the 90-days prior to index procedure,
16. Subject has undergone a percutaneous procedure of 8F sheath or less using a suture mediated closure device or manual/mechanical pressure for haemostasis in the target vessel, within the 30-days prior to index procedure,
17. History of DVT or pulmonary embolism or venous thrombotic event,
18. Splenectomy or suffering psoriasis or paraesthesia of the ipsilateral leg,
19. Further planned endovascular/catheter-based procedure in the target leg in the 30-days following the index procedure,
20. Subject is enrolled in another investigational medical device or drug study,
21. Subject has been previously enrolled in this clinical study,
22. Subject is unable to maintain ipsilateral leg still during the index procedure (restless leg syndrome),
23. Current COVID-19 infection (with or without symptoms), recent positive test for COVID-19 within two weeks, or recent exposure to a person with COVID-19 infection within two weeks.

    Procedural Exclusion Criteria:
24. Anatomically the common femoral vein is substantially posterior to the femoral artery, confirmed by Duplex ultrasound,
25. Initial common femoral venous access achieved other than with the use of an ultrasound guided access approach,
26. If the venous access is, or suspected of being, via an artery,
27. Difficult dilation during initial target femoral vein access (e.g., that damages or kinks dilators) while step-dilating up to the large-bore device,
28. During venous puncture, the target femoral vein suspected to have experienced a posterior venous wall needle puncture or underwent > one needle puncture during the primary procedure, with a needle larger than a micropuncture needle (> 21 gauge or > 0.819 mm diameter). (Note: not an exclusion if micropuncture technique under ultrasound guidance used for femoral vein access [Ref. 30, 31]),
29. Subject has a tissue tract (i.e., estimated distance from skin entry point to venous anterior surface at venotomy) expected to be greater than 8 cm,
30. Significant blood loss requiring transfusion of blood products during primary procedure or within 30-days prior to index procedure,
31. Activated clotting time (ACT) > 250 seconds immediately prior to sheath removal or if ACT measurements are expected to be > 250 seconds for more than 24 hours after index procedure,
32. Target puncture site is in a vascular graft,
33. Target venotomy greater than 26F,
34. Target femoral vein diameter is less than 7 mm, based on Duplex ultrasound or angiography,
35. Evidence of venous diameter stenosis > 20% within 15 mm proximal or distal to venotomy site based on Duplex ultrasound or angiography,
36. Target venotomy has been made in the superficial femoral vein, profunda femoris vein (deep femoral vein), great saphenous vein or located less than 15 mm distal (cranial) to the bifurcation of either the profunda femoris or great saphenous vein and common femoral vein,
37. Target venotomy located behind (posterior) or above (cranial) to the inguinal ligament based upon bony landmarks (above femoral head on A-P projection),
38. Subjects with an acute haematoma > 4 cm diameter, arteriovenous fistula, pseudoaneurysm or intraluminal thrombosis at the target access site identified intra-procedurally,
39. Evidence of bleeding around the primary procedure sheath (VARC type 1/BARC type 2 or higher),
40. Intra-procedural (angiographic or Duplex ultrasound) evidence of venous laceration, dissection or stenosis within the femoral vein that would preclude use of the PerQseal Elite device,

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint- Combined rate of both Major and Minor access site complications | through 30 Days
  the combined rate of both Major and Minor access site complications attributable to the PerQseal Elite device§ through 30-days, as adjudicated by the Clinical Events Committee (CEC) as study device related.
Primary Effectiveness Endpoint - Time to Haemostasis | 20 Minutes
  Time to Haemostasis (TTH) defined as elapsed time in minutes from PerQseal Elite (Introducer-sheath and Delivery-device) removal to first observed cessation of common femoral vein (CFV) bleeding (clinically acceptable cessation of venous bleeding), excluding cutaneous or subcutaneous oozing, and in the absence of a developing haematoma. This is assessed at the end of the index procedure prior leaving the operating room/catheterisation laboratory.

SECONDARY OUTCOMES:
Secondary Effectiveness Endpoint - PerQseal Elite Technical Success Rate | 10 Minutes
  PerQseal Elite Technical Success Rate is defined as the number of PerQseal Elite devices that are deployed and achieve haemostasis (i.e., cessation of venous bleeding excluding cutaneous or subcutaneous oozing) without need for more than 10 minutes of firm, adjunctive manual compression or alternative treatment (other than adjunctive endovascular ballooning) at target access site, divided by the total number of PerQseal Elite devices where deployment was attempted.
Secondary Effectiveness Endpoint - PerQseal Elite Treatment Success Rate | through 30 days
  PerQseal Elite Treatment Success Rate is defined as the number of subjects who meet PerQseal Elite Technical Success without experiencing a device related Access Site Complication (based on CEC adjudication) through 30-days, divided by the total number of subjects where PerQseal Elite device deployment was attempted.
Secondary Effectiveness Endpoint -Time to Device Deployment (TTDD) | 20 Minutes
  Time to Device Deployment is defined as the time from insertion of the PerQseal Elite delivery device into the PerQseal Elite Introducer sheath to complete removal of the PerQseal Elite (delivery device and introducer-sheath) from the subject following PerQseal Elite deployment.
Secondary Effectiveness Endpoint - Time to Ambulation | through 24 hours
  Time to Ambulation is defined as: the elapsed time from PerQseal Elite removal from the subject post deployment until the subject can walk 20 feet/6 meters without venous re-bleeding at the target access site. This endpoint will be evaluated only for subjects who are ambulatory (e.g., not confined to wheelchair or bed) at the time of enrolment.
Secondary Effectiveness Endpoint - Total Closure Time | 40 Minutes
  Total Closure Time is defined as: Time to Haemostasis (TTH) plus Time to Device Deployment (TTDD).

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus UMC, Rotterdam, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No